CLINICAL TRIAL: NCT04649788
Title: Prospective Randomized Comparison of Efficacy and Safety of Ultrasound-guided Axillary Vein Access Versus Cephalic Venous Cutdown for Implantation of Cardiac Electronic Devices
Brief Title: Ultrasound-guided Axillary Vein Access Versus Cephalic Venous Cutdown for Implantation of Cardiac Electronic Devices.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL19_0540; ANSM (Other: 2019-A02952-55)
Record Dates: First submitted 2020-10-15; First posted 2020-12-02 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2023-02

CONDITIONS: Pacemaker; Implantable Cardioverter-defibrillator
Keywords: pacemaker; implantable cardioverter-defibrillator; axillary vein; cephalic vein; ultrasound

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-guided axillary vein access (Active Comparator): This group of patients will receive the cardiac implantable electronic device with ultrasound-guided axillary venous access.
  Interventions: Device: Ultrasound-guided axillary vein access
- Cephalic vein access (Active Comparator): This group of patients will receive the cardiac implantable electronic device with cephalic venous access.
  Interventions: Device: Cephalic vein access

INTERVENTIONS:
Device: Ultrasound-guided axillary vein access — Venous access is performed through ultrasound-guided axillary vein puncture and Seldinger technique. After venous access is obtained, a guide-wire is advanced through the access needle, and the tip of the guide-wire is positioned in the right cardiac atrium.
  Arms: Ultrasound-guided axillary vein access
Device: Cephalic vein access — Venous access is performed through a cephalic vein cutdown approach. After venous access is obtained, a guide-wire is advanced and the tip of the guide-wire is positioned in the right cardiac atrium.
  Arms: Cephalic vein access

SUMMARY:
Venous access is a fundamental step in lead insertion for endovenous cardiac implantable electronic devices (CIED). Cephalic vein cutdown is the most widely used technique in Europe. Ultrasound-guided axillary vein access is a promising alternative but there is a lack of clinical evidence supporting this technique.

The purpose of this study is to compare the efficacy and safety of ultrasound-guided axillary vein access versus cephalic venous cutdown for implantation of endovenous CIED.

Half of patients is implanted using an ultrasound-guided axillary vein puncture. The other half is implanted using a cephalic vein cutdown. After venous access is achieved, implantation procedure is identical in the two arms.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Indication for endovenous pacemaker or cardioverter-defibrillator (single or double room)

Exclusion Criteria:

* History of previously implanted endocardial lead
* Indication for cardiac resynchronization therapy
* Impossibility of venous access
* Unable/unwilling to provide informed consent
* Pregnant or breastfeeding woman
* Participating in another clinical study which can interfere with this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
Success of venous access | Intervention time (day 0)
  This outcome is measured by the operator during the intervention. It is the ability to successfully cannulate the vein and have all needed guidewire in the right atrium using the assigned venous access technique.
  The outcome is a binary value: success or failure.

SECONDARY OUTCOMES:
Time to venous access | Intervention time (day 0)
  Time from cutaneous incision to reach the right atrium with all needed guidewire using the assigned venous access technique
Procedure duration | Intervention time (day 0)
  Time from cutaneous incision to skin suture
Fluoroscopy time | Intervention time (day 0)
  Duration of fluoroscopy use during intervention
X-Ray exposure | Intervention time (day 0)
  X-ray exposure during intervention, measured in mGycm2
Complication | Intervention time (day 0)
  All implant related complications including brachial plexus palsy, major pocket hematoma (hematoma requiring evacuation or transfusion or prolonged hospitalization), pneumothorax, hemothorax, pericardial effusion, lead dislodgement, device infection, venous thrombosis.
Cardiac implantable electronic device (CIED) related infection | Month 3
  Local and systemic signs of CIED related infection will be monitored during follow-up. The definition and classification of CIED related infection are based on the current guideline and expert consensus statement.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon - Hopital de la Croix Rousse, Lyon, France

REFERENCES:
- [Result] Charles P, Ditac G, Montoy M, Thenard T, Courand PY, Lantelme P, Harbaoui B, Fareh S. Intra-pocket ultrasound-guided axillary vein puncture vs. cephalic vein cutdown for cardiac electronic device implantation: the ACCESS trial. Eur Heart J. 2023 Dec 7;44(46):4847-4858. doi: 10.1093/eurheartj/ehad629. PMID 37832512